CLINICAL TRIAL: NCT05799521
Title: A Novel Nasal Treatment for COVID-19
Brief Title: A Nasal Treatment for COVID-19
Acronym: COVD-TX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, James F. Chmiel, Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15989
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: COVID-19; Healthy
MeSH Terms: conditions — COVID-19 | interventions — Optate; Glycine; Saline Solution

STUDY DESIGN:
Intervention Model Description: The study model arms will include participants with COVID-19 receiving treatment (experimental type), participants with COVID-19 receiving placebo (placebo comparator type), healthy controls receiving treatment (experimental type), and healthy controls receiving placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Providing pharmacy will randomize doses and provide blinded doses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Participants with COVID-19:Treatment (Experimental): Participants with COVID-19:Treatment - subjects on this treatment arm will receive study drug
  Interventions: Drug: Optate
- Participants with COVID-19: Placebo (Placebo Comparator): Participants with COVID-19: Placebo - subjects on this arm will get placebo
  Interventions: Drug: Placebo
- Healthy Controls: Treatment (Experimental): Healthy Controls: Treatment - subjects on this treatment arm will receive study drug
  Interventions: Drug: Optate
- Healthy Controls: Placebo (Placebo Comparator): Healthy Controls: Placebo - subjects on this arm will get placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Optate — Alkaline Buffer
  Other Names: Glycine
  Arms: Healthy Controls: Treatment; Participants with COVID-19:Treatment
Drug: Placebo — Normal Saline
  Other Names: Normal Saline
  Arms: Healthy Controls: Placebo; Participants with COVID-19: Placebo

SUMMARY:
The goal of this study is to test an investigational new inhaled medication called Optate.

DETAILED DESCRIPTION:
The goal of this study is to test an investigational new inhaled medication called Optate. Investigational means it has not been approved by the Food and Drug Administration (FDA) for this use. The investigators hypothesize that Optate will reduce the length of symptoms and disease severity in patients with COVID-19 (Coronavirus disease of 2019) through inhibition of SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2) viral replication within the upper and lower airways. Testing this hypothesis is important because treatments for COVID-19 are needed alongside vaccines. COVID-19 begins in the nasal passages, so targeted therapies to the nasal passages at early stages of the disease may prevent severe disease from occurring.

ELIGIBILITY:
COVID-19 PARTICIPANTS Inclusion Criteria: Subjects, 18 and above, with mild COVID-19 upper respiratory tract infection symptoms

* positive rapid COVID-19 test
* Ordinal Scale for Clinical Improvement < 3 (OSCI, Appendix 2) and/or
* Fever > 100 degree F and/or
* Nasal congestion

Exclusion Criteria:

* FEV1 (Forced Exhaled Volume) < 55% predicted on the day of study procedures
* OSCI ≥ 3 (Objective Structured Clinical Exam)
* Pregnancy
* Inability to follow commands or perform study procedures including spirometry, coordinated inhalation of study medication

HEALTHY CONTROLS Inclusion Criteria: Subjects, 18 and above, without mild COVID-19 upper respiratory tract infection symptoms

* negative rapid COVID-19 test
* No known medical problems or taking any medication that, in the investigator's opinion, would make them unsuitable for participation.

Exclusion Criteria:

* Pregnancy
* Inability to follow commands or perform study procedures including spirometry, coordinated inhalation of study medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in SARS-CoV-2 Levels | Immediately before and one-hour after treatment
  SARS-CoV-2 levels will be measured in nasal wash before and one hour after Optate or placebo administration
Change in SNOT-22 score | Immediately before and one-hour after treatment
  SNOT-22 scores (a validated, 22-item quality of life instrument survey) will be assessed immediately prior to Optate or placebo administration. The SNOT-22 assesses five domains (nasal, ear/facial, sleep, function and emotion) on a Likert scale from 0-5, where 0 means no problems and 5 means the worst possible problems. The total score ranges from 0-110, with higher scores indicating more severe symptoms. Scores will be reassessed one hour after administration.
Change in SNOT-22 score | Immediately before and 24-hours after treatment
  SNOT-22 scores (a validated, 22-item quality of life instrument survey) will be assessed immediately prior to Optate or placebo administration. The SNOT-22 assesses five domains (nasal, ear/facial, sleep, function and emotion) on a Likert scale from 0-5, where 0 means no problems and 5 means the worst possible problems. The total score ranges from 0-110, with higher scores indicating more severe symptoms. Scores will be reassessed 24 hours after administration.

SECONDARY OUTCOMES:
Change in SARS-CoV-2 Levels | Immediately before and one-hour after treatment
  SARS-CoV-2 levels will be measured in exhaled breath condensate before and one hour after Optate or placebo administration
Change in nasal pH | Immediately before, immediately after and one-hour after treatment
  Nasal pH will be measured by a nasal pH meter before, immediately after and one hour after Optate or placebo administration

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Davis MD, Donn SM, Ward RM. Administration of Inhaled Pulmonary Vasodilators to the Mechanically Ventilated Neonatal Patient. Paediatr Drugs. 2017 Jun;19(3):183-192. doi: 10.1007/s40272-017-0221-9. PMID 28374138
- [Background] Davis MD, Hunt J. Exhaled breath condensate pH assays. Immunol Allergy Clin North Am. 2012 Aug;32(3):377-86. doi: 10.1016/j.iac.2012.06.003. Epub 2012 Jul 10. PMID 22877616
- [Background] Davis MD, Walsh BK, Dwyer ST, Combs C, Vehse N, Paget-Brown A, Pajewski T, Hunt JF. Safety of an alkalinizing buffer designed for inhaled medications in humans. Respir Care. 2013 Jul;58(7):1226-32. doi: 10.4187/respcare.01753. Epub 2012 Dec 18. PMID 23258576
- [Background] Hunt JF, Fang K, Malik R, Snyder A, Malhotra N, Platts-Mills TA, Gaston B. Endogenous airway acidification. Implications for asthma pathophysiology. Am J Respir Crit Care Med. 2000 Mar;161(3 Pt 1):694-9. doi: 10.1164/ajrccm.161.3.9911005. PMID 10712309
- [Background] Ngamtrakulpanit L, Yu Y, Adjei A, Amoah G, Gaston B, Hunt J. Identification of Intrinsic Airway Acidification in Pulmonary Tuberculosis. Glob J Health Sci. 2010 Apr;2(1):106-110. doi: 10.5539/gjhs.v2n1p106. PMID 21197384
- [Background] Ricciardolo FL, Gaston B, Hunt J. Acid stress in the pathology of asthma. J Allergy Clin Immunol. 2004 Apr;113(4):610-9. doi: 10.1016/j.jaci.2003.12.034. PMID 15100663
- [Background] Shin HW, Shelley DA, Henderson EM, Fitzpatrick A, Gaston B, George SC. Airway nitric oxide release is reduced after PBS inhalation in asthma. J Appl Physiol (1985). 2007 Mar;102(3):1028-33. doi: 10.1152/japplphysiol.01012.2006. Epub 2006 Nov 16. PMID 17110506
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] Paget-Brown AO, Ngamtrakulpanit L, Smith A, Bunyan D, Hom S, Nguyen A, Hunt JF. Normative data for pH of exhaled breath condensate. Chest. 2006 Feb;129(2):426-430. doi: 10.1378/chest.129.2.426. PMID 16478862